CLINICAL TRIAL: NCT00146471
Title: Efficacy and Safety of Levetiracetam in the Inpatient Treatment of Alcohol Withdrawal Syndrome [Sicherheit Und Wirksamkeit Von Levetiracetam (Keppra) für Die Behandlung Des stationären Alkoholentzugsyndroms]
Brief Title: Efficacy and Safety of Levetiracetam in the Inpatient Treatment of Alcohol Withdrawal Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Martin Schaefer, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kep-F10.3.01
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2008-09

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: alcohol withdrawal; detoxification; Inpatients; alcohol dependence according to DSM-IV/ICD-10; withdrawal symptoms
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Levetiracetam
- 1: Diazepam plus Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — 1500-2000 mg daily add-on or Placebo Diazepam as needed
  Other Names: KEPPRA
  Arms: 2
Drug: Placebo — 1500-2000 mg daily add-on or Placebo Diazepam as needed
  Arms: 1: Diazepam plus Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of levetiracetam for treating alcohol withdrawal syndrome (AWS) in inpatients (vs. placebo). The primary come-out parameter is the reduction of the total needed amount of diazepam for add-on treatment of acute alcohol withdrawal symptoms. The secondary come-out parameter are - safety criteria (AE) - reduction of alcohol withdrawal score over the days.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18-65 years.
* Meets criteria for alcohol dependence according to DSM-IV/ICD-10
* Known withdrawal symptoms in the past in case of discontinuation of alcohol consumption
* Hospital admission for alcohol detoxification
* Able to provide a written informed consent.
* Able to follow verbal and written instructions (incl. a sufficient knowledge of German language).
* Must be medically acceptable for study treatment. No past or present physical disorder that is likely to deteriorate during participation. No ECG abnormality which would likely worsen during participation and no clinical laboratory abnormality that would also suggest deterioration during treatment.
* Have a negative urine drug screen for benzodiazepines or heroine or methadone

Exclusion Criteria:

* Current diagnosis of any other substance dependence syndrome other than alcohol dependence (excluding nicotine and caffeine dependence).
* History of idiopathic epilepsy.
* Patient with any current clinically significant psychiatric disorder (acute suiciality) or developmental disorder (including organic mental disorder), like psychotic disorders.
* Patients with the following complications of alcoholism (lifetime): acute delirium tremens, hallucinatory alcoholic state, Korsakoff's syndrome, Wernicke encephalopathy, decomposed liver cirrhosis (Child B, C), suspected cirrhosis with the following clinical symptoms detected at clinical exam: signs of portal hypertension and signs of hepato-cellular failure, thrombocytopenia.
* Subjects with known sensitivity of previous adverse reaction to levetiracetam
* Contra-indication (hypersensitivity to levetiracetam or pyrrolidone derivatives) or known non-response to levetiracetam.
* History of severe GI disease which might render absorption of the medication difficult or produce medical instability of the patient which would include active peptic ulcer disease, ulcerative colitis, regional colitis, or evidence by history or physical exam of GI bleeding.
* Patients with any clinically significant acute or chronic progressive neurological, gastrointestinal, cardiovascular, hepatic, renal, haematological, endocrine, dermatological or respiratory disease, such as diabetes, severe infection, acute alcoholic hepatitis, or any other medical condition with significant worsening of the clinical situation of the patient that might interfere with the evaluation of study medication.
* Female patients pregnant, breast-feeding or of child bearing age and not protected by effective contraceptive such as implants, injectables, combined oral contraceptives, some IUDS, sexual abstinence, sterilization or vasectomized partner.
* Actually continuous use of pharmacological agents that are known to lower the seizure threshold or augment or decrease the alcohol withdrawal syndrome.
* Subjects with known sensitivity of previous adverse reaction to diazepam or clonidine
* Contra-indication or known non-response to diazepam or clonidine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of levetiracetam for treating alcohol withdrawal syndrome in inpatients. The primary come-out parameter is the reduction of the amount of diazepam for add-on treatment of acute alcohol withdrawal | during trial

SECONDARY OUTCOMES:
Secondary come-out parameters are - safety criteria (AE) - reduction of alcohol withdrawal score over the days | during trial

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Charité Campus Mitte, Klinik für Psychiatrie und Psychotherapie
Locations (5):
- Germany (5):
  - MLU Halle-Wittenberg, Halle, Sachen/Anhalt
  - Charité - Universitätsmedizin Berlin, Campus Charité Mitte, Klinik für Psychiatrie und Psychotherapie, Berlin, State of Berlin
  - Psychiatrische Klinik der Charité im St.-Hedwig Krankenhaus, Berlin, State of Berlin
  - Klinik für Psychiatrie und Suchtmedizin, Kliniken Essen Mitte, Essen
  - Zentrum für Seelische Gesundheit, Rhede

REFERENCES:
- [Background] Krebs M, Leopold K, Richter C, Kienast T, Hinzpeter A, Heinz A, Schaefer M. Levetiracetam for the treatment of alcohol withdrawal syndrome: an open-label pilot trial. J Clin Psychopharmacol. 2006 Jun;26(3):347-9. doi: 10.1097/01.jcp.0000219926.49799.89. No abstract available. PMID 16702910
- [Derived] Richter C, Hinzpeter A, Schmidt F, Kienast T, Preuss UW, Plenge T, Heinz A, Schaefer M. Levetiracetam for the treatment of alcohol withdrawal syndrome: a multicenter, prospective, randomized, placebo-controlled trial. J Clin Psychopharmacol. 2010 Dec;30(6):720-5. doi: 10.1097/jcp.0b013e3181faf53e. PMID 21105289